CLINICAL TRIAL: NCT02236182
Title: A Double-blind, Placebo Controlled Trial to Assess the Safety of Two-week Administration of 80 mcg q.i.d. and 160 mcg q.i.d. of Ipratropium Bromide, as Delivered by the RESPIMAT® Device, in Patients With Chronic Obstructive Pulmonary Disease
Brief Title: Study to Assess the Safety of Ipratropium Bromide, in Patients With Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 244.2489
Record Dates: First submitted 2014-09-09; First posted 2014-09-10 (Estimated); Last update posted 2014-09-12 (Estimated); Status verified 2014-09

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Ipratropium

ARMS (3):
- Ipratropium Bromide low (Experimental): delivered via RESPIMAT®
  Interventions: Drug: Ipratropium Bromide low dose
- Ipratropium Bromide high (Experimental): delivered via RESPIMAT®
  Interventions: Drug: Ipratropium Bromide high dose
- Placebo (Placebo Comparator): delivered via RESPIMAT®
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ipratropium Bromide low dose
  Arms: Ipratropium Bromide low
Drug: Placebo
  Arms: Placebo
Drug: Ipratropium Bromide high dose
  Arms: Ipratropium Bromide high

SUMMARY:
Study to assess the safety of two-week administration of 80 and 160 mcg of ipratropium bromide as delivered by the RESPIMAT® device and as determined by 24 hours ambulatory ECG monitoring in COPD patients. To assess the overall safety of the two doses of ipratropium bromide as delivered by the RESPIMAT® device when administered over a two-week period.

ELIGIBILITY:
Inclusion Criteria:

All patients must have a diagnosis of COPD and must meet the following spirometric criteria:

* Patients must have relatively stable, moderate to severe airway obstruction with an FEV1 <=65% of predicted normal and FEV1 <=70% of forced vital capacity (FVC). Predicted normal value will be calculated according to Morris

  * Males: FEV1 = 0.093 (Height in inches)-0.032 (age)-1.343
  * Females: FEV1 = 0.085 (Height. in inches)-0.025(age)-1.692
* Male or female patients 40 years of age or older
* Patients must have a smoking history of more than 10 pack-years. A pack-year is defined as the equivalent of smoking one pack of 20 cigarettes per day for a year
* Patients must be able to perform pulmonary function tests (PFTs) and maintain records during the study period as required in the protocol
* Patients must be able to be trained in the proper use of an inhalation aerosol and the RESPIMAT™ device
* Patients must have a baseline electrocardiogram (ECG) with no clinical relevant arrhythmias or conduction system disease (e.g. right or left bundle branch block, second degree AV block or higher)
* Patients must have an oxygen saturation of >=90% for >=92% of the recording time on overnight oximetry
* All patients must sign an Informed Consent Form prior to participation in the trial (i.e., at least 24 hours (h) prior to the screening visit (Visit 1))

Exclusion Criteria:

* Patients with clinically relevant diseases other than COPD will be excluded. A clinically relevant disease is defined as a disease which in the opinion of the investigator may either put the patient at risk because of participation in the study or a disease with may influence the results of the study or patient's ability to participate in the study
* Patients with a recent history (i.e. one year or less) of myocardial infarction
* Patients with a recent history (i.e. one year or less) of heart failure or patients with any past history or active cardiac arrhythmia requiring drug therapy
* Patients who have a pacemaker
* Patients with clinically relevant abnormal baseline hematology, blood chemistry or urinalysis. If the abnormality defines a disease listed as an exclusion criterion the patient is excluded
* All patients with serum glutamic oxaloacetic transaminase / Aspartate aminotransferase (SGOT/AST) >80 IU/L, serum glutamic pyruvic transaminase / Alanine transaminase (SGPT/ALT) >80 IU/L, bilirubin >2.0 mg/dl, or creatinine >2.0 mg/dl will be excluded regardless of the clinical condition. Repeat laboratory evaluation will be not be conducted in these subjects
* Patients who have a blood eosinophil count >=600/mm3. A Repeat eosinophil count will be not be conducted in these patients
* Patients with a history of cancer, other than treated basal cell carcinoma, within the last 5 years
* Patients with a history of life-threatening pulmonary obstruction, or a history of cystic fibrosis or bronchiectasis
* Patients who have undergone thoracotomy with pulmonary resection. Patients with a history of thoracotomy for other reason should be evaluated per exclusion criterion No. 1
* Patients with a history of asthma, allergic rhinitis or atopy
* Patients with a history of and/or active alcohol or drug abuse
* Patients with known active tuberculosis
* Patients with an upper respiratory tract infection or COPD exacerbation in the past 6 weeks prior to the screening visit (Visit 1) or during the baseline period
* Patients with known symptomatic prostatic hypertrophy or bladder neck obstruction
* Patients with known narrow-angle glaucoma
* Patients with current significant psychiatric disorders
* Patients with regular use of daytime oxygen therapy
* Patients who are being treated with cromolyn sodium or nedocromil sodium
* Patients who are being treated with antihistamines
* Patients using oral corticosteroid medication at unstable doses (i.e. less than six weeks on a stable dose) or at a dose in excess of the equivalent of 10 mg of prednisone per day or 20 mg every other day
* Patients who are being treated with beta-blocker medication
* Patients who have had changes in their therapeutic plan within the last six weeks prior to the screening visit (visit 1)
* Pregnant or nursing women or women of childbearing potential not using a medically approved means of contraception (e.g., oral contraceptive, intrauterine devices, diaphragm or Norplant®)
* Patients with known hypersensitivity to ant cholinergic drugs or any other components of the ATROVENT® RESPIMAT™ solution including bacteriostatic agent benzalkonium chlorid (BAC) and edetic acid (EDTA)
* Patients who have taken an investigational drug within 1 month or 6 half-lives (whichever is longer) prior to the screening visit (visit1)
* Previous participation in this study

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 1998-07; Primary Completion 1999-02 (Actual)

PRIMARY OUTCOMES:
Assessment of clinical significant findings in 24-hour ambulatory ECG monitoring | Pre-treatment, on Day 7 and 13
Number of patients with adverse events | Up to 15 days after first drug administration
Number of patients with clinical significant findings in ECG | Up to 15 days after first drug administration
Number of patients with clinical significant findings in vital signs | Up to 15 days after first drug administration
Number of patients with clinical significant findings in laboratory tests | Up to day 15 after drug administration
Number of patients with paradoxical bronchospasm | Up to 15 days after first drug administration

SECONDARY OUTCOMES:
FEV1 (forced expiratory volume in the first second) AUC0-4 (Area under the curve from 0 to 4 hours) | Pre-treatment, up to 4 h after drug administration on Day 1 and 14
Peak FEV1 | On Day 1 and 14
Onset of therapeutic FEV1 response | On Day 1 and 14
Time to peak FEV1 response | On Day 1 and 14
AUC(0-6h) (Area under the plasma concentration-time curve from 0 to 6 h) | Day 14
Cmax (maximum plasma concentration) | Day 14
Cmin(0h) (minimum plasma concentration before inhalation) | Day 14
Cmin(6h) (minimum plasma concentration at 6 hours after inhalation) | Day 14
Ae(0-2h) (urine excretion between 0 to 2 h) | Day 14
Ae(0-6h) (urine excretion between 0 to 6 h) | Day 14